CLINICAL TRIAL: NCT00625456
Title: A Phase I Dose Escalation Study of JX-594 (Thymidine Kinase-deleted Vaccinia Virus Plus GM-CSF) Administered by Intravenous Infusion in Patients With Refractory Solid Tumors
Brief Title: Safety Study of Recombinant Vaccinia Virus to Treat Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Organization: SillaJen, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX594-IV-011
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2012-03

CONDITIONS: Melanoma; Lung Cancer; Renal Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck
Keywords: phase I; advanced metastatic solid tumors; oncolytic virus; vaccinia virus; melanoma; lung cancer; renal cell carcinoma; squamous cell carcinoma of the head and neck; Pexa-Vec
MeSH Terms: conditions — Melanoma; Lung Neoplasms; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck; Vaccinia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm, dose escalation (Experimental): dose escalation starting dose 1e5 pfu/kg bw to 3e7 pfu/kg bw; Recombinant Vaccinia GM-CSF (JX-594)
  Interventions: Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)

INTERVENTIONS:
Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594) — Intravenous Dosage from 1 x 10^5 pfu/kg to 3 x 10^7 pfu/kg Intravenous infusion is administered once over a 60 minute period
  Other Names: JX-594

SUMMARY:
This is a Phase I, open-label, dose-escalation trial in patients with advanced/metastatic solid tumors refractory to standard therapy; tumors may include malignant melanoma, non-small cell lung cancer, renal cell carcinoma, and squamous cell carcinoma of the head and neck. These tumor types were selected because evidence of biological activity was observed in these tumor types in a Phase I study of JX-594 (Pexa-Vec) administered by intratumoral injection in patients with metastatic disease to the liver. Patients will receive treatment at one of five dose levels in a sequential dose-escalating design.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, advanced/metastatic solid tumor refractory to standard therapy or the patient has refused or does not tolerate the standard therapy; tumors may include malignant melanoma, non-small cell lung cancer, renal cell carcinoma, and squamous cell carcinoma of the head and neck
* At least one measurable tumor mass by CT/MRI (i.e. lesion that can accurately be measured in at least one dimension with longest diameter > 1 cm)
* At least one tumor mass amenable to biopsy and/or FNA
* Expected survival for approximately 16 weeks or longer
* Karnofsky Performance Score (KPS) ≥ 70
* Age ≥18 years
* WBC ≥ 3,500 cells/mm3 and ≤ 50,000 cells/mm3
* ANC ≥ 1,500 cells/mm3
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100,000 plts/mm3
* Total bilirubin ≤ 1.5 x ULN
* AST, ALT ≤ 2.5 x ULN
* Serum chemistries within normal limits (WNL) or Grade 1 - If patients are diabetic or have a screening random glucose > 160 mg/dL, a fasting glucose must be done and patients must be WNL or Grade 1 in order to be eligible for the study.
* Acceptable coagulation status: INR ≤ (ULN + 10%)
* CD4 count ≥ 500/mm3

Exclusion Criteria:

* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids)
* Known myeloproliferative disorders requiring systemic therapy
* History of exfoliative skin condition (e.g. eczema or ectopic dermatitis) requiring systemic therapy
* Tumor(s) invading a major vascular structure (e.g. carotid artery)
* Tumor(s) in location that would potentially result in significant clinical adverse effects if post-treatment tumor swelling were to occur (e.g. tumors impinging on the upper airway or affecting biliary tract drainage, etc.)
* Clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions
* Severe or unstable cardiac disease
* Current, known CNS malignancy (history of completely resected or irradiated brain metastases allowed)
* Received anti-cancer therapy within 4 weeks prior to first treatment (6 weeks in case of mitomycin C or nitrosoureas)
* Use of anti-viral, anti-platelet, or anti-coagulation medication [Patients who discontinue such medications within 7 days prior to first treatment may be eligible for this study.]
* Pulse oximetry O2 saturation <90% at rest
* Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination

Household contact exclusions:

* Women who are pregnant or nursing an infant
* Children < 5 years old
* History of exfoliative skin condition (e.g. eczema) that at some stage has required systemic therapy
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximally-tolerated dose (MTD) and/or maximum-feasible dose (MFD) of JX-594 administered by intravenous (IV) infusion | 4 weeks
Safety/Toxicity: Incidence of treatment-related adverse events; treatment-related serious adverse events; treatment-related Grade 3/4 toxicities; and clinically-significant, treatment-related changes from baseline in routine laboratory parameters | 4 weeks

SECONDARY OUTCOMES:
Determine the JX-594 pharmacokinetics and pharmacodynamics over time following IV infusion | 4 weeks
Determine the immune response to JX-594 following IV infusion | 4 weeks
Determine the delivery of JX-594 to, and concentration within, solid tumors following IV infusion | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Kirn, MD, Study Director — Jennerex Inc.
Locations (4):
- United States (3):
  - Billings Clinic, Billings, Montana
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
- Ottawa Health Research Institute, Ottawa, Ontario, Canada